CLINICAL TRIAL: NCT02040636
Title: Safety and Immunogenicity of Tetanus and Diphtheria Toxoids Adsorbed Combined With Component Pertussis Vaccine and Inactivated Poliomyelitis Vaccine (TdcP-IPV) Compared to Tetanus and Diphtheria Toxoids Adsorbed Combined With Component Pertussis Vaccine and Inactivated Poliomyelitis Vaccine (TdcP-IPV) and Hepatitis B Vaccine Given Concurrently In Adolescents 11-14 Years of Age
Brief Title: Study of Tetanus and Diphtheria Toxoids Adsorbed Combined With Component Pertussis Vaccine and Inactivated Poliomyelitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TD9809
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Pertussis; Tetanus; Diphtheria; Poliomyelitis; Hepatitis B
Keywords: Pertussis; Tetanus; Diphtheria; Poliomyelitis; Hepatitis B; Acellular Pertussis Vaccines
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria; Poliomyelitis; Hepatitis B | interventions — Tetanus Toxoid; Poliovirus Vaccine, Inactivated; Hepatitis B Vaccines; Recombivax HB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental): Participants randomized to receive Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and Inactivated Poliomyelitis Vaccine (TdcP-IPV) at month 0, Hepatitis B at months 1, 2 and 7.
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and IPV; Biological: Hepatitis B vaccine
- Study Group 2 (Active Comparator): Participants randomized to receive Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and Inactivated Poliomyelitis Vaccine (TdcP-IPV) + Hepatitis B at month 0, Hepatitis B at months 1 and 6.
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and IPV; Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and IPV — 0.5 mL, Intramuscular
  Other Names: TdcP-IPV
Biological: Hepatitis B vaccine — 0.5 ml, Intramuscular
  Other Names: Recombivax HB®

SUMMARY:
Primary objective:

* To determine the safety and immunogenicity of tetanus and diphtheria toxoids adsorbed combined with component pertussis and inactivated poliomyelitis vaccine grown on vero cells (TdcP-IPV) compared to tetanus and diphtheria toxoids adsorbed combined with component pertussis and inactivated poliomyelitis vaccine grown on vero cells (TdcP-IPV) and Hepatitis B vaccine administered concurrently in adolescents 11-14 years of age.

Secondary objective:

* To determine whether concurrent administration of TdcP-IPV and Hepatitis B vaccines at 11-14 years of age results in detectable immunologic interactions between components of the two vaccines.

DETAILED DESCRIPTION:
Participants will be randomized into one of 2 groups to receive either a dose of the TdcP-IPV on Day 0 (visit 1) and Hepatitis B vaccine on subsequent visits 2, 3 and 4 (Group 1); or no vaccination on Day 0, concomitant administration of TdcP-IPV and Hepatitis B vaccine on Day 28 (Visit 2) and Hepatitis B vaccine on subsequent visits 3 and 4 (Group 2).

All participants will be followed up for immunogenicity and safety

ELIGIBILITY:
Inclusion Criteria:

* Age 11 years and < 14 years of age.
* Signed, witnessed and dated informed consent that is obtained prior to the first study intervention.
* Judged to be in good health on the basis of reported medical history.
* Plans to remain in the study area for the length of the trial.
* All minors have a parent or legal guardian who can read, write and understand English or French.
* Pregnancy test to be performed on all female participants at the time of enrollment into the study (prior to day of first immunization visit).

Exclusion Criteria:

* Pregnancy.
* Known or suspected primary disease of the immune system [conditions suspected of having an immunologic component such as autoimmune diseases (rheumatoid arthritis or inflammatory bowel disease) will not be excluded unless they meet exclusion criterion 3 or are sufficiently clinically active to meet exclusion criterion 5].
* Malignancy or is receiving immunosuppressive therapy (e.g., daily systemic prednisone ≥ 1 mg/kg would be excluded, participants who are taking topical and inhaled steroids could be included in the study as could participants on a "short course" of oral steroids, 5-7 days, as long as there are not two courses within the previous two week period).
* Prior receipt of any pertussis, diphtheria, tetanus or polio containing vaccines, including Hepatitis B vaccine, within the past 5 years.
* Any significant underlying chronic disease, including malignancy, cardiopulmonary disease, renal or hepatic dysfunction.
* Known impairment of neurologic function or seizure disorder of any etiology.
* Personal history of physician diagnosed or laboratory confirmed pertussis disease within the last 2 years.
* Receipt of blood products or immunoglobulin within the previous 3 months.
* Known or suspected allergy to any of the vaccines intended for use in the study or any of the vaccine components including neomycin, streptomycin and polymyxin B.
* Receipt of any vaccine within 2 weeks of receiving a study vaccine.
* Daily use of non-steroidal anti-inflammatory drugs.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 277 (Actual)
Dates: Start 1999-01; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Seroprotection against diphtheria and tetanus antigens after vaccination with either Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and Inactivated Poliomyelitis (Tdcp-IPV) or concurrent Tdcp-IPV and Hepatitis B vaccine | Day 0 (pre-vaccination) and 1 month, 3, 5 and 10 years post-vaccination
  Seroprotection defined as: Diphtheria levels ≥ 0.01 IU/mL and ≥ 0.1 IU/mL; Tetanus levels ≥ 0.01 EU/mL and ≥ 0.1 EU/mL.
Geometric Mean Titers for Diphtheria and Tetanus after vaccination with either Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine & Inactivated Poliomyelitis Vaccine (Tdcp-IPV) or concurrent Tdcp IPV and Hepatitis B vaccine | Day 0 (pre-vaccination) and 1 month, 3, 5 and 10 years post-vaccination
  Diphtheria antibodies assayed using enzyme-linked immunoassay; Tetanus antibodies were assessed using microneutralization assay
Number of participants reporting solicited injection site reactions, solicited systemic reactions, unsolicited adverse events, and serious adverse events occurring during trial | Day 0 up to day 30 following each vaccination
  Solicited local injection site reactions: Redness, Swelling, and Tenderness. Solicited systemic reactions: Altered Appetite, Headache, General Malaise, Nausea, Vomiting and Muscle aches.

SECONDARY OUTCOMES:
Geometric Mean Titers for Pertussis antibodies after vaccination with either Tetanus and Diphtheria Toxoids Adsorbed Combined with Component Pertussis Vaccine and Inactivated Poliomyelitis Vaccine (TdcP IPV) or concurrent Tdcp IPV and Hepatitis B vaccine | Day 0 (pre-vaccination) and 1 month, 3, 5 and 10 years post-vaccination
  Anti pertussis toxoid, anti filamentous hemagglutinin, anti fimbriae 2 + 3 and anti Pertactin antibodies were assayed by enzyme linked immunoassay; Polio types 1, 2, and 3 were assayed using neutralizing antibodies to poliovirus types1, 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Ltd.
Locations (1):
- Winnipeg, Manitoba, Canada

REFERENCES:
- [Result] Embree J, Law B, Voloshen T, Tomovici A. Immunogenicity, safety, and antibody persistence at 3, 5, and 10 years postvaccination in adolescents randomized to booster immunization with a combined tetanus, diphtheria, 5-component acellular pertussis, and inactivated poliomyelitis vaccine administered with a hepatitis B virus vaccine concurrently or 1 month apart. Clin Vaccine Immunol. 2015 Mar;22(3):282-90. doi: 10.1128/CVI.00682-14. Epub 2014 Dec 24. PMID 25540274
- See also: Related Info — http://www.sanofipasteur.com